CLINICAL TRIAL: NCT01800357
Title: Efficacy and Safety of Mildronate for Acute Ischemic Stroke: Study Protocol for a Randomized, Double-blind, Placebo-controlled Phase II Multicenter Trial
Brief Title: Efficacy and Safety of Mildronate for Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xijing-007
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-01

CONDITIONS: Acute Ischemic Stroke
Keywords: randomized trial; acute ischemic stroke; mildronate
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mildronate (Experimental): infusion of mildronate
  Interventions: Drug: infusion of mildronate; Drug: aspirin
- placebo (Placebo Comparator): infusion of placebo mildronate
  Interventions: Drug: placebo; Drug: aspirin

INTERVENTIONS:
Drug: infusion of mildronate — infusion of mildronate(500mg) once a day and for 14 days
  Arms: mildronate
Drug: placebo — infusion of plabcebo once a day and for 14 days
  Arms: placebo
Drug: aspirin — infusion of aspirin (100mg) once a day for days

SUMMARY:
This study seeks to evaluate the efficacy and safety of mildronate injection in treating acute ischemic stroke

DETAILED DESCRIPTION:
a randomized, double-blind, placebo-controlled phase II multicenter trial is conducted to evaluate the efficacy and safety of mildronate injection in patients with acute ischemic stroke. patients will be randomized to receive a 14-day treatment of placebo or mildronate (500mg/5ml/each).Primary end-point is the modified Rankin scale at 3 monthes. Secondary end-point is the NIHSS scores and the Barthel index at 8 days and 15days. The safety end-point is defined as the incidence of adverse events, the change of Samples for routine laboratory tests and vital signs. Analysis is by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

- have a clinical diagnosis of acute ischemic stroke have CT or MRI brain imaging NIHSS scores:5~22 on the first stage

Exclusion Criteria:

- have other intracranial pathologies are pregnant or nursing have significant drug or alcohol misuse have been in a clinical trial in the past 3 months are unlikely to be available for follow-up have been given thrombolytic therapy or medication forbidden by study protocol have a neurological or psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
the modified Rankin scale | 3 months

SECONDARY OUTCOMES:
NIHSS scores | 8 days
NIHSS scores | 15 days
the Barthel index | 8 days
the Barthel index | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital; Yi Zhu, MD, Study Chair — the Department of Neurology , Xijing Hospital
Locations (1):
- the Department of Neurology , Xijing Hospital, Xi'an, Shaanxi, China